CLINICAL TRIAL: NCT03571542
Title: Evaluation of the Respiratory Function in Renal Transplanted Children : a Prospective, Multicenter French Study
Brief Title: Evaluation of the Respiratory Function in Renal Transplanted Children
Acronym: SPIROKID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Collaborators: Lille University Hospital (Unknown); Hospices Civils de Lyon (Other); NECKER UNIVERSITY HOSPITAL (Unknown); Hopital Universitaire Robert-Debre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC18_0142
Record Dates: First submitted 2018-05-31; First posted 2018-06-27 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Respiratory Tract Disease; Kidney Transplantation; Pediatric
Keywords: Children; transplanted; kidney transplantation; respiratory function; pulmonary function tests; respiratory disease; immunosuppression
MeSH Terms: conditions — Respiratory Tract Diseases; Respiratory Aspiration; Respiration Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: pulmonary function — The aim of this study is to assess the respiratory function thanks to pulmonary function tests in renal transplanted children in France.

SUMMARY:
Objectives:

While a respiratory abnormality was found in 50% of pediatric renal transplant recipients in a study conducted in Belgium and the Netherlands in 2008, the respiratory status of transplanted children in France remains unknown. The primary objective of this study is to assess the prevalence of respiratory impairment and its characteristics in children with renal transplant. The secondary objective is to study its association with some potential risk factors such as immunosuppressive therapy or humoral immunodeficiency.

Methodology:

This interventional study aims to recruit the 385 children currently being followed by 5 French pediatric renal transplant centers between June 2018 and November 2019. A clinical and functional respiratory assessment will be carried out during the routine annual follow-up of the transplant recipient. Children with clinical signs of concern or abnormal spirometry will be referred to a respiratory specialist. Pharmacokinetic assays of immunosuppressant therapy and the exploration of humoral function will also be performed. The prevalence and type of respiratory abnormalities will be described. Logistic regression will be used to explore the association between potential risk factors and impaired respiratory function.

Expected results:

This study will be the first to evaluate the respiratory status of children with renal transplants in France. The prospective, multi- centered nature of the study, in addition to the large cohort size (which represents two thirds of children with renal transplants in France) will guarantee current, reliable, and representative data for the target population. We will provide new knowledge by precisely characterizing the type of lung injury and looking for potential risk factors. If our study confirms the high prevalence of pulmonary impairment in children with renal transplants, systematic monitoring of respiratory function may be recommended to enable early diagnosis and management. The expected individual and public health benefits would be significant by limiting the appearance of long-term, irreversible sequelae (such as non-cystic-fibrosis bronchiectasis) and improving the quality of life of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplanted
* Patients of 2 to 20 years old
* Followed in one the five centers mentionned above (Nantes, Necker, Robert Debré, Lyon, Lille)

Exclusion Criteria:

* Disaggrement from the patient and/or his/her legal representant
* Impossibility to do the pulmonary function test
* Cystic fibrosis
* Patient with another transplant (heart, lung, liver)

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 385 (Estimated)
Dates: Start 2018-07-16 (Actual); Primary Completion 2022-07-16 (Estimated); Study Completion 2022-07-16 (Estimated)

PRIMARY OUTCOMES:
Respiratory alteration | at the inclusion
  An alteration of the pulmonary function tests (PFT) values or the presence of chronic respiratory symptoms/treatment (questionnaire)

SECONDARY OUTCOMES:
risk factors linked to an alteration of the respiratory function | at the inclusion
  We will analyse the relation between several exposure variables or the potential risk factors (medical past, medication, infectious diseases,...) and the presence of an alteration of the respiratory function.
  Clinical datas will be gathered thanks to a questionnaire on the medical past and the respiratory state of the child.
  The usual biological measures will be done at the annual check up (exploring immunity, pharmacological dosages, renal function, for example).

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHRU Lille, Lille
  - Hospices Civiles de Lyon, Lyon
  - CHU de Nantes, Nantes
  - Hôpital Universitaire Necker Enfants Malades, Paris
  - Robert Debre Hospital, Paris